CLINICAL TRIAL: NCT05859334
Title: A Phase 2 Study of Erdafitinib in Patients With Recurrent or Progressive IDH-Wild Type Glioma With an FGFR-TACC Gene Fusion
Brief Title: Testing the Anti-cancer Drug Erdafitinib for Brain Cancers That Have Returned or Progressed Following Treatment
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2023-03776; NCI-2023-03776 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10559 (Other: University Health Network Princess Margaret Cancer Center LAO); 10559 (Other: CTEP); UM1CA186644 (NIH)
Record Dates: First submitted 2023-05-13; First posted 2023-05-16 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Glioma; Recurrent WHO Grade 2 Glioma; Recurrent WHO Grade 3 Glioma; Recurrent WHO Grade 4 Glioma
MeSH Terms: conditions — Glioma | interventions — Specimen Handling; erdafitinib; Magnetic Resonance Spectroscopy; Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (erdafitinib) (Experimental): Patients receive erdafitinib PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo MRI, OCT, and collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Drug: Erdafitinib; Procedure: Magnetic Resonance Imaging; Procedure: Optical Coherence Tomography

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Erdafitinib — Given PO
  Other Names: Balversa; JNJ 42756493; JNJ-42756493; JNJ42756493
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Optical Coherence Tomography — Undergo OCT
  Other Names: OCT; Optical Coherence Tomography (OCT)

SUMMARY:
This phase II trial tests how well erdafitinib works in controlling IDH-wild type (WT), FGFR-TACC gene fusion positive gliomas that have come back after a period of improvement (recurrent) or that are growing, spreading, or getting worse (progressive). Erdafitinib is in a class of medications called kinase inhibitors. It works by blocking the action of an abnormal FGFR protein that signals tumor cells to multiply. This may help keep tumor cells from growing and may kill them. Giving erdafitinib may help to slow the growth of, or to shrink, tumor cells in patients with recurrent or progressive IDH-wild type gliomas with FGFR-TACC gene fusion.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the preliminary anti-tumor activity of erdafitinib in patients with recurrent or progressive IDH-WT glioma with FGFR-TACC gene fusion as measured by the best response at any time during treatment in terms of objective response rate (ORR).

SECONDARY OBJECTIVES:

I. To determine the safety and tolerability of erdafitinib in patients with recurrent or progressive IDH-WT glioma with FGFR-TACC gene fusion.

II. To assess the overall survival (OS) of erdafitinib in patients with recurrent or progressive IDH-WT glioma with FGFR-TACC gene fusion.

III. To assess the progression free survival (PFS) at 6 months of patient with IDH-WT glioma with FGFR-TACC gene fusion treated with erdafitinib.

OUTLINE: This is a dose-escalation study of erdafitinib followed by a dose-expansion study.

Patients receive erdafitinib orally (PO) once daily (QD) on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo magnetic resonance imaging (MRI), optical coherence tomography (OCT), and collection of blood samples throughout the trial.

After study completion, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be >= 18 years of age
* Patient must have histologically confirmed IDH-WT gliomas (grade 2-4) as per World Health Organization (WHO) 2016 or 2021 classification
* Tumor tissue should be positive for FGFR-TACC gene fusion as per any local next generation sequencing (NGS) (Clinical Laboratory Improvement Act [CLIA]-approved) assay described in background section
* The disease should be recurrent or progressive glioma after initial anti-tumor treatment with at least 1 line of treatment including surgical resection, radiation therapy and/or chemotherapy
* For patients with WHO grade 3 or 4 glioma and progressive disease < 12 weeks after completion of chemoradiotherapy, progression can be defined by the following set of criteria:

  * New enhancement outside of the radiation field (beyond the high-dose region or 80% isodose line)
  * If there is unequivocal evidence of viable tumor on histopathologic sampling (e.g., solid tumor areas. i.e., > 70% tumor cell nuclei in areas), high or progressive increase in Ki-67 proliferation index compared with prior biopsy, or evidence for histologic progression or increased anaplasia in tumor)
* For patients with WHO grade 3 or 4 glioma and progressive disease >= 12 weeks after completion of chemoradiotherapy, progression can be defined by the following set of criteria:

  * New contrast-enhancing lesion outside of radiation field on decreasing, stable, or increasing doses of corticosteroids
  * Increase by >= 25% in the sum of the products of perpendicular diameters between the first post-radiotherapy scan, or a subsequent scan with smaller tumor size, and the scan at 12 weeks or later on stable or increasing doses of corticosteroids
  * For patients receiving antiangiogenic therapy, significant increase in T2/fluid attenuated inversion recovery (FLAIR) non-enhancing lesion may also be considered progressive disease. The increased T2/FLAIR must have occurred with the patient on stable or increasing doses of corticosteroids compared with baseline scan or best response after initiation of therapy and not be a result of comorbid events (e.g., effects of radiation therapy, demyelination, ischemic injury, infection, seizures, postoperative changes, or other treatment effects)
* For patients with WHO grade 2 glioma progression is defined by any one of the following:

  * Development of new lesions or increase of enhancement (radiological evidence of malignant transformation)
  * A 25% increase of the T2 or FLAIR non-enhancing lesion on stable or increasing doses of corticosteroids compared with baseline scan or best response after initiation of therapy, not attributable to radiation effect or to comorbid events
* There must be measurable disease (enhancing or non-enhancing as per Response Assessment in Neuro-Oncology [RANO] or RANO-low-grade glioma [LGG] criteria), as evaluated on pre-treatment MRI
* Patient understands the procedures and investigational nature of the study drug and agrees to comply with study requirements by providing written informed consent
* Patient must have Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (or Karnofsky >= 60%)
* Absolute neutrophil count >= 1000/uL
* Hemoglobin > 8 g/dL (Patients are allowed to be transfused to this level)
* Platelets >= 100 x 10^9/L
* Serum total bilirubin =< 1.5 x upper limit of normal (ULN), unless considered due to Gilbert's disease or disease involvement following approval by the medical monitor
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 3 x institutional ULN
* Creatinine clearance > 30 mL/min (patients with mild or moderate renal impairment) based on the Cockroft-Gault glomerular filtration rate (GFR) estimation
* Patient must have normal serum phosphate level as per local laboratory parameters. (Medical management allowed)
* Patient must be recovered from any clinically relevant toxic effects of any prior surgery, radiotherapy, or chemotherapy treatment with temozolomide
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients should be New York Heart Association Functional Classification class 2B or better
* The effects of erdafitinib on the developing human fetus are unknown. For this reason and because FGFR inhibitors are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and one month after completion of erdafitinib administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and one month after completion of erdafitinib administration
* Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants

Exclusion Criteria:

* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to erdafitinib
* Patients requiring any medications or substances that are moderate CYP2C9 inducers and strong CYP3A4 inducers are ineligible. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Patients with uncontrolled intercurrent illness
* Pregnant women are excluded from this study because erdafitinib is an FGFR inhibitor agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with erdafitinib, breastfeeding should be discontinued if the mother is treated with erdafitinib
* Current central serous retinopathy (CSR) or retinal pigment epithelial detachment of any grade
* Corrected QT interval (QTc) prolongation as confirmed by electrocardiography (ECG) at screening (Fridericia; QTc > 480 milliseconds)
* Patients who have previously received FGFR inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-01-04 (Actual); Primary Completion 2026-10-23 (Estimated); Study Completion 2026-10-23 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Up to 2 years
  Defined as the proportion of patients with either complete response or partial response as per Response Assessment in Neuro-Oncology criteria. The response rate will be estimated along with the corresponding 95% confidence interval using the binomial exact method. Univariable and multivariable logistic regression models will be used to estimate the associations between study covariates and response status. Odds ratios and corresponding 95% confidence intervals and p-values will be reported.

SECONDARY OUTCOMES:
Incidence of dose-limiting toxicities | Up to 28 days
  Analyzed based on National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Incidence of adverse events (AEs) and serious AEs | Up to 2 years
  Analyzed based on NCI CTCAE version 5.0.
Progression-free survival | Time between date of enrollment and date of progression or date of death from any cause, assessed at 6 months
  Kaplan-Meier method will be used to estimate survival rates for pre-specified time points along with 95% confidence intervals. Hazard ratios (HRs) will be estimated using Cox proportional hazards regression model to examine the associations of study covariates with time-to-event outcomes along with corresponding 95% confidence intervals and p-values if these are estimable.
Overall survival | Time between the date of enrollment and date of death from any cause, censored at the last date of follow-up, assessed up to 2 years
  Kaplan-Meier method will be used to estimate survival rates for pre-specified time points along with 95% confidence intervals. HRs will be estimated using Cox proportional hazards regression model to examine the associations of study covariates with time-to-event outcomes along with corresponding 95% confidence intervals and p-values if these are estimable.

CONTACTS AND LOCATIONS:
Overall Officials: Macarena I De La Fuente, Principal Investigator — University Health Network Princess Margaret Cancer Center LAO
Locations (27):
- United States (27):
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Memorial Hospital East, Shiloh, Illinois
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm